CLINICAL TRIAL: NCT01119612
Title: Prenatal Iron Supplements: Safety and Efficacy in Tanzania
Acronym: MAL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD061232
Record Dates: First submitted 2010-04-30; First posted 2010-05-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Malaria; Anemia
Keywords: Malaria; Iron; Pregnancy; Anemia; Birth Weight
MeSH Terms: conditions — Malaria; Anemia; Birth Weight | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron (Active Comparator)
  Interventions: Dietary Supplement: Iron
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Iron — Daily oral dose of 60 mg from enrollment until delivery
  Arms: Iron
Other: Placebo — Daily oral dose from enrollment until delivery
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety and efficacy of prenatal iron supplementation in an area of high malaria burden among women who are not anemic or iron deficient.

DETAILED DESCRIPTION:
Iron deficiency anemia and malaria are urgent public health problems in sub-Saharan Africa, including Tanzania. There is a paucity of good quality randomized trials assessing the safety and efficacy of iron supplementation in pregnancy, and its effects on perinatal health outcomes. Prenatal iron supplementation is recommended based on its demonstrated benefit in preventing and treating maternal anemia. There is limited data on the efficacy of iron supplementation on pregnancy outcomes, including birth weight. There are also concerns regarding the use of iron supplementation, particularly among non-anemic women. In particular, there is a lack of research on the safety and efficacy of prenatal iron supplementation in developing regions, characterized by extensive burden of iron deficiency, malaria, and other endemic infectious diseases. Evidence from randomized controlled trials is urgently needed to examine the safety and efficacy of iron supplements among pregnant women in malaria endemic regions, particularly among women who are not anemic.

NOTE: The time frames listed for the maternal malaria and hemoglobin outcomes were updated on 4/22/15. This record initially indicated that maternal malaria anemia and hemoglobin would be measured at several specific time points throughout the study. Instead, maternal malaria was measured throughout pregnancy and hemoglobin was measured only at delivery. Due to an oversight, we did not update this record when this protocol change took effect at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* at or before 27 weeks of gestation
* primigravida or secundigravidae
* not anemic (defined as Hb<8.5 g/dL)
* not iron deficient (defined as serum ferritin <12 μg/L)
* HIV-uninfected
* intend to stay in Dar es Salaam until delivery and for at least six weeks thereafter.

Exclusion Criteria:

* After 27 weeks gestation
* not primigravida or secundigravidae
* anemic
* iron deficient
* HIV-infected
* High iron stores at baseline (i.e., serum ferritin >200 μg/L)
* do not intend to stay in Dar es Salaam until delivery and for at least six weeks thereafter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of placental malaria | Delivery
  Placental infection status will be categorized as infected if there are asexual parasites in the placenta blood; not infected if the placental blood smear is negative; or status unknown if no placental smear is available.
Placental malaria parasite density | Delivery
  Placental malaria parasite density will be defined as number of parasites per μL of blood or 200 white blood cells; the latter will be converted to a count per μL of blood assuming a count of 8000 WBC/μL.
Infant birth weight | Delivery
  Continuous measurement
Maternal hemoglobin | Delivery
  Continuous measurement

SECONDARY OUTCOMES:
Low birth weight | Delivery
  Low birth weight will be defined as birth weight less than 2500 grams.
Maternal malaria infection | During pregnancy
  Maternal malaria will be defined as fever within the last 72 hours with any parasitemia on a peripheral blood smear.
Maternal anemia | Delivery
  Anemia will be defined as hemoglobin less than 11 g/dl. Severe anemia will be defined as less than 8.5 g/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Zul Premji, MD, MSC, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health And Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Finkelstein JL, Cuthbert A, Weeks J, Venkatramanan S, Larvie DY, De-Regil LM, Garcia-Casal MN. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD004736. doi: 10.1002/14651858.CD004736.pub6. PMID 39145520
- [Derived] Abioye AI, Hughes MD, Sudfeld CR, Premji Z, Aboud S, Hamer DH, Roberts DJ, Duggan CP, Fawzi WW. The effect of iron supplementation on maternal iron deficiency anemia does not differ by baseline anemia type among Tanzanian pregnant women without severe iron deficiency anemia. Eur J Nutr. 2023 Mar;62(2):987-1001. doi: 10.1007/s00394-022-03029-0. Epub 2022 Nov 8. PMID 36344770
- [Derived] Yang J, Wang M, Tobias DK, Rich-Edwards JW, Darling AM, Abioye AI, Pembe AB, Madzorera I, Fawzi WW. Gestational weight gain during the second and third trimesters and adverse pregnancy outcomes, results from a prospective pregnancy cohort in urban Tanzania. Reprod Health. 2022 Jun 16;19(1):140. doi: 10.1186/s12978-022-01441-7. PMID 35710384
- [Derived] Yang J, Wang D, Darling AM, Liu E, Perumal N, Fawzi WW, Wang M. Methodological approaches to imputing early-pregnancy weight based on weight measures collected during pregnancy. BMC Med Res Methodol. 2021 Feb 5;21(1):24. doi: 10.1186/s12874-021-01210-3. PMID 33546607
- [Derived] Etheredge AJ, Premji Z, Gunaratna NS, Abioye AI, Aboud S, Duggan C, Mongi R, Meloney L, Spiegelman D, Roberts D, Hamer DH, Fawzi WW. Iron Supplementation in Iron-Replete and Nonanemic Pregnant Women in Tanzania: A Randomized Clinical Trial. JAMA Pediatr. 2015 Oct;169(10):947-55. doi: 10.1001/jamapediatrics.2015.1480. PMID 26280534